CLINICAL TRIAL: NCT01050946
Title: Phase II Study: HSCT Using CD34 Selected Mismatched Related Donor and One Umbilical Cord Unit
Brief Title: Hematopoietic Stem Cell Transplantation (HSCT) Using CD34 Selected Mismatched Related Donor and One Umbilical Cord Unit
Acronym: Haplo/Cord
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Only one patient was enrolled. Due to low accrual study was terminated
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Parameswaran Hari, Professor of Medicine, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCW 11491
Record Dates: First submitted 2010-01-14; First posted 2010-01-18 (Estimated); Results first posted 2015-09-25 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Leukemia, Lymphocytic, Acute; Leukemia, Lymphocytic, Chronic; Leukemia, Myelocytic, Acute; Leukemia, Myeloid, Chronic; Lymphoma, Non-Hodgkin; Lymphoma, Hodgkins
Keywords: Unrelated Umbilical Cord Blood Transplant(UCB); CD34+ Selected mismatched related donor; Haploidentical donor; hematopoietic stem cell transplantation(HSCT); ALL; Leukemia, Lymphocytic, Acute; AML; Leukemia, Myelocytic, Acute; CML; Leukemia, Myeloid, Chronic; NHL; Lymphoma, Non-Hodgkin; HL; Lymphoma, Hodgkins
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Non-Hodgkin; Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Haploidentical/cord transplant (Other): Haploidentical/cord transplant with the precondition regimen at discretion of treating physician.
  Interventions: Biological: Haploidentical/cord transplant

INTERVENTIONS:
Biological: Haploidentical/cord transplant — Myeloablative preparative regimen of chemotherapy and radiation followed by mismatch related(haploidentical)donor and one unit umbilical cord blood transplantation.
  Conditioning Regimens Choice of regimen at the discretion of the treating physician
  1. Fludarabine 30mg/m2(Days-7,-6,-5,-4,-3)-,Melphalan 70mg/m2(Day -3,-2), ATG 1.5mg/m2(Day-7,-5,-3,-1)
  2. Fludarabine 50mg/m2(Day -6,-5,-4,-3,-2),Busulfan 3.2mg/kg(Day -5,-4,-3,-2),400cGY Total Body Irradiation(TBI)Day-1,ATG 1.5mg/kg(Day-7,-5,-3,-1)
  Day 0 -Haploidentical donor and one umbilical cord blood unit infusion
  Other Names: Cord Blood Transplant

SUMMARY:
This study is a means of providing transplantation to those patients who would be a stem cell transplant candidate who do not have an appropriate donor.

The use of CD34 selected haploidentical donor with an umbilical cord unit may help provide earlier engraftment without the need for long term immunosuppression.

This study tests a new method of bone marrow transplantation called combined haploidentical-cord blood transplantation. In this procedure, some of the blood forming cells (the stem cells) from a partially human leukocyte antigen (HLA) matched (haploidentical) related donor are collected from the blood, as well as cells from an umbilical cord are transplanted into the patient (the recipient) after administration of a "conditioning regimen". A conditioning regimen consists of chemotherapy and sometimes radiation to the entire body (total body irradiation, or TBI), which is meant to destroy the cancer cells and suppress the recipient's immune system to allow the transplanted cells to take (grow).

DETAILED DESCRIPTION:
This method of stem cell transplantation is designed to overcome some of the limitations of other alternative donor transplant options. Use of unrelated umbilical cord unit (UCB) donors appears to allow a greater degree of HLA mismatch with acceptable rates of GVHD. However, when UCB transplant was studied in the adult population, investigators discovered several limitations. One major limitation with UCB was delayed engraftment, resulting in higher risk of infection in the early post transplant period. The limitations to cord blood transplant involve delayed engraftment resulting in early complications such as infections. The main limitation associated with haploidentical donors is the significant immunosuppression required to prevent/treat aGVHD. Use of this combined modality of transplantation appears to allow for rapid neutrophil engraftment from the haploidentical donor and coupled with long term hematopoiesis from the UCB donor, thus requiring less long term immunosuppression.

This study tests a new method of bone marrow transplantation called combined haploidentical-cord blood transplantation. In this procedure, some of the blood forming cells (the stem cells) from a partially HLA matched (haploidentical) related donor are collected from the blood, as well as cells from an umbilical cord are transplanted into the patient (the recipient) after administration of a "conditioning regimen". A conditioning regimen consists of chemotherapy and sometimes radiation to the entire body (total body irradiation, or TBI),

One of two 'conditioning regimens' which will be determined by the physician.

1. FLUDARABINE, MELPHALAN, ATG

   Fludarabine 30mg/m2(Days-7,-6,-5,-4,-3)-,Melphalan 70mg/m2(Day -3,-2), ATG 1.5mg/m2(Day-7,-5,-3,-1)
2. FLUDARABINE, BUSULFAN, 400 CGY TBI, ATG Fludarabine 50mg/m2(Day -6,-5,-4,-3,-2),Busulfan 3.2mg/kg(Day -5,-4,-3,-2) 400cGY Total Body Irradiation(TBI)Day-1,ATG 1.5mg/kg(Day-7,-5,-3,-1)

Day 0 -Haploidentical donor and one umbilical cord blood unit infusion

Filgrastim will be administered daily from day +1 until blood counts have completely recovered. Tacrolimus and another immunosuppressant, Cellcept, starting before transplant also to reduce the risks of graft versus host disease and to promote the growth of the graft. Tacrolimus will be given daily from two days before the transplant until at least three months after transplantation. Cellcept, will be tapered after the cells engraft.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 65 years old
* Patient has a related family member(haploidentical) or unrelated which is 5 of 10 HLA identical match.

Standard Risk

* Acute myelogenous leukemia: CR1 with high risk cytogenetics or molecular abnormalities such as FLT-3 ITD, or CR2 with a first remission that must have lasted > 1 year.
* Acute Lymphocytic Leukemia: CR1, in order to be standard risk must NOT have Philadelphia Chromosome.
* Chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL): Must be refractory to fludarabine or fail to have a complete or partial response after therapy with a regimen containing fludarabine (or another nucleoside analog, e.g. 2-CDA, pentostatin) or experience disease relapse within 12 months after completing therapy with a regimen containing fludarabine (or another nucleoside analog).
* Chronic myelogenous leukemia: resistant to or intolerant of TKI, in CP1 or CP2, or with a mutation that suggests resistance to TKI.
* Myelodysplastic Syndrome: RA, RARS, must be IPSS ≥ INT-2, Blasts <5%.

High Risk Patients:

* Acute myelogenous leukemia: Patients with CR2 are considered high risk if they have high risk cytogenetics, or molecular abnormalities or CR1 lasted for less than 1 year. Any evidence of active disease or no blasts in an acellular marrow.
* Acute Lymphocytic Leukemia: CR1- with Ph+ disease, CR2/+ with any cytogenetics. Any evidence of active disease.
* Chronic myelogenous leukemia- CP2/+, AP1/+, resistant or intolerant to TKI.
* Hodgkin's or Non Hodgkin's lymphoma- Disease recurrence following an autologous transplant, or high risk disease not thought to benefit from autologous transplant.
* Chronic lymphocytic leukemia- that is resistant to fludarabine, and never has been in remission or with stable disease/progressive disease
* Multiple myeloma: Must have had prior treatment. Patients in CR2 or greater can be considered, must have already failed autologous transplant Previous autologous transplant,must have been greater than 6 months prior to undergoing this transplant.
* Myelodysplastic syndrome: RAEB
* Other Myeloproliferative disorders including myelofibrosis, spent phase p Vera,Essential thrombocytosis,CMML.

Exclusion Criteria:

* Patients <18 years old Disease related criteria
* APML, presence of t(15,17) in first CR
* Patients with good risk AML, for example t(8;21), or inv 16, or normal cytogenetics with FLT-3-ITD negative, NPM-1 positive disease in 1st CR
* MDS IPSS < INT-2 Miscellaneous Criteria
* Recipients who have a matched related sibling or unrelated donor
* If recipient has evidence of anti-HLA antibodies directed against cord or haplo-donor as determined byflowPRA.

Underlying health criteria:

* Zubrod performance status > 2 (see Appendix E)
* Life expectancy is limited to less than 8 weeks by concomitant illness
* Patients with severely decreased LVEF (EF < 40%)
* Impaired pulmonary function tests (PFT's) (FVC, FEV1, DLCO < 45% predicted)
* Estimated Creatinine Clearance <50 ml/min
* Serum bilirubin> 2.0 mg/dl or SGPT >3 x upper limit of normal
* Evidence of chronic active hepatitis or cirrhosis
* HIV-positive
* Patient is pregnant
* Patient or guardian not able to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Palmer, M.D., Principal Investigator — Medical College of Wisconsin

REFERENCES:
- [Derived] van Besien K, Artz A, Champlin RE, Guarneri D, Bishop MR, Chen J, Gergis U, Shore T, Liu H, Rondon G, Mayer SA, Srour SA, Stock W, Ciurea SO. Haploidentical vs haplo-cord transplant in adults under 60 years receiving fludarabine and melphalan conditioning. Blood Adv. 2019 Jun 25;3(12):1858-1867. doi: 10.1182/bloodadvances.2019000200. PMID 31217161

RESULTS

PARTICIPANT FLOW:
Recruitment Details: FDA approval was granted on 6/18/11 and went into effect on 7/18/11.Recruitment period started from the 7/18/11 until study closure on 3/28/13, All recruitment took place in the clinic setting. Only one patient was accrued.
Groups:
- Haploidentical/Cord Transplant: Haploidentical/cord transplant with the preconditioning regimen at discretion of treating physician.
  Haploidentical/cord transplant : Myeloablative preparative regimen of chemotherapy and radiation followed by mismatch related(haploidentical)donor and one unit umbilical cord blood transplantation.
  Conditioning Regimens Choice of regimen at the discretion of the treating physician
  1. Fludarabine 30mg/m2(Days-7,-6,-5,-4,-3)-,Melphalan 70mg/m2(Day -3,-2), ATG 1.5mg/m2(Day-7,-5,-3,-1)
  2. Fludarabine 50mg/m2(Day -6,-5,-4,-3,-2),Busulfan 3.2mg/kg(Day -5,-4,-3,-2),400cGY Total Body Irradiation(TBI)Day-1,ATG 1.5mg/kg(Day-7,-5,-3,-1)
  Day 0 -Haploidentical donor and one umbilical cord blood unit infusion
Period: Overall Study
Arm/Group | Haploidentical/Cord Transplant
Started | 1
Completed | 1 (Patient signed consent 2/3/2011. Patient had their transplant 2/15/2011. Patient died 9/2/2011)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Haploidentical/Cord Transplant: Haploidentical/cord transplant with the precondition regimen at discretion of treating physician.
  Haploidentical/cord transplant : Myeloablative preparative regimen of chemotherapy and radiation followed by mismatch related(haploidentical)donor and one unit umbilical cord blood transplantation.
  Conditioning Regimens Choice of regimen at the discretion of the treating physician
  1. Fludarabine 30mg/m2(Days-7,-6,-5,-4,-3)-,Melphalan 70mg/m2(Day -3,-2), ATG 1.5mg/m2(Day-7,-5,-3,-1)
  2. Fludarabine 50mg/m2(Day -6,-5,-4,-3,-2),Busulfan 3.2mg/kg(Day -5,-4,-3,-2),400cGY Total Body Irradiation(TBI)Day-1,ATG 1.5mg/kg(Day-7,-5,-3,-1)
  Day 0 -Haploidentical donor and one umbilical cord blood unit infusion
Arm/Group | Haploidentical/Cord Transplant
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective is to Estimate the Overall Survival, Separately in the Two Risk Strata.
Time Frame: 3 years
Population: Only one patient enrolled on study. Patient died prior to time frame of 3 years. It is not possible to assess this outcome measure.
Groups:
- Haploidentical/Cord Transplant: Haploidentical/cord transplant with the precondition regimen at discretion of treating physician.
  Haploidentical/cord transplant: Myeloablative preparative regimen of chemotherapy and radiation followed by mismatch related(haploidentical)donor and one unit umbilical cord blood transplantation.
  Conditioning Regimens Choice of regimen at the discretion of the treating physician
  1. Fludarabine 30mg/m2(Days-7,-6,-5,-4,-3)-,Melphalan 70mg/m2(Day -3,-2), ATG 1.5mg/m2(Day-7,-5,-3,-1)
  2. Fludarabine 50mg/m2(Day -6,-5,-4,-3,-2),Busulfan 3.2mg/kg(Day -5,-4,-3,-2),400cGY Total Body Irradiation(TBI)Day-1,ATG 1.5mg/kg(Day-7,-5,-3,-1)
  Day 0 -Haploidentical donor and one umbilical cord blood unit infusion
Arm/Group | Haploidentical/Cord Transplant
Number analyzed (Participants) | 0

2. Secondary Outcome: Time to Relapse: To Assess the Incidence of Acute Leukemia or Lymphoma Relapse From Day of Transplant
Description: NOT analyzed since there was only patient and no relapse was observed till patient passed away
Time Frame: 2 years
Population: Patient did not live to 2 years, no relapse observed
Arm/Group | Haploidentical/Cord Transplant
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to Neutrophil Engraftment: To Assess the Incidence of Neutrophil Engraftment From Day of Transplant
Description: time to neutrophil recovery after transplant
Time Frame: 100 days
Population: Patient engrafted neutrophils and platelets but no statistical analysis possible
Arm/Group | Haploidentical/Cord Transplant
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Platelet Engraftment: To Assess the Incidence of Platelet Engraftment From Day of Transplant,
Time Frame: 100 days
Population: No further analysis reported as only one patient enrolled
Arm/Group | Haploidentical/Cord Transplant
Number analyzed (Participants) | 0

5. Secondary Outcome: Time to Acute GVHD: We Will Assess the Incidence and Severity of Grades II-IV and Grades III-IV Acute GVHD From Day of Transplant.
Time Frame: 100 days
Population: only one participant - no analysis done
Arm/Group | Haploidentical/Cord Transplant
Number analyzed (Participants) | 0

6. Secondary Outcome: Transplant Related Mortality (TRM): TRM is Death Occurring in Patients in Continuous Complete Remission.
Time Frame: 1 year
Population: only pt who was enrolled died of TRM
Measure: Number; unit: participants
Arm/Group | Haploidentical/Cord Transplant
Number analyzed (Participants) | 1
participants | 1

7. Secondary Outcome: Disease-free Survival:Death or Relapse Will be Considered Events for This Endpoint.
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Haploidentical/Cord Transplant
Number analyzed (Participants) | 1
participants | 0

ADVERSE EVENTS:
Time Frame: From the time the patient signed consent until the patient's death.
Arm/Group | Haploidentical/Cord Transplant
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Haploidentical/Cord Transplant (N=1)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Patient underwent an EGD on 5/5/11 to evaluate for GI motility problems and gastric outlet obstruction. During the procedure patient became hypoxic and required intubation. Patient developed Acute Respiratory Distress Syndrome (ARDS).
Acute Renal Injury (Renal and urinary disorders) | 1 (1) — Acute Renal Injury with previous history of tubular necrosis on 3/29/11.
Confusion (Psychiatric disorders) | 1 (1) — Patient was admitted to hospital for management of altered mental status for acute onset of confusion.
Death (Infections and infestations) | 1 (1) — Due to worsening CMV and BK virus/ Hemorrhagic Cystitis patient decided to receive only palliative care. Patient was receiving palliative care at the time of her death.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Haploidentical/Cord Transplant (N=1)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Patient underwent an EGD on 5/5/11 to evaluate for GI motility problems and gastric outlet obstruction. During the procedure patient became hypoxic and required intubation. Patient developed Acute Respiratory Distress Syndrome (ARDS).
Acute Renal Injury (Renal and urinary disorders) | 1 (1) — Acute Renal Injury with previous history of tubular necrosis on 3/29/11.
Confusion (Psychiatric disorders) | 1 (1) — Patient was admitted to hospital for management of altered mental status for acute onset of confusion.
Death (Infections and infestations) | 1 (1) — Due to worsening CMV and BK virus/ Hemorrhagic Cystitis patient decided to receive only palliative care. Patient was receiving palliative care at the time of her death.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes